CLINICAL TRIAL: NCT03667521
Title: Prospective Cross-sectional Study on the Prevalence of Stool Outlet Obstruction After Laparoscopic Sacrocolpopexie at the KSA
Brief Title: Prevalence of Stool Outlet Obstruction After Laparoscopic Sacrocolpopexie
Status: Completed | Type: Observational
Sponsor: Kantonsspital Aarau (Other)
Responsible Party: Principal Investigator, Dimitri Sarlos, Head of the Womens Hospital Kantonsspital Aarau, chief of gynecology and gyn. oncology, head of the breast and gyn. tumor center, Kantonsspital Aarau
Other Study IDs: SACRO-GYN-KSA
Record Dates: First submitted 2018-09-10; First posted 2018-09-12 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Stool Outlet Obstruction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- non-nerve-sparing laparaoscopic sacrocolpopexy.
- nerve-sparing laparaoscopic sacrocolpopexy.
  Interventions: Procedure: nerve-sparing laparaoscopic sacrocolpopexy

INTERVENTIONS:
Procedure: nerve-sparing laparaoscopic sacrocolpopexy — nerve-sparing laparaoscopic sacrocolpopexy implemented after 2010
  Groups: nerve-sparing laparaoscopic sacrocolpopexy.

SUMMARY:
The aim was to evaluate the prevalence of stool outlet obstruction after laparoscopic sacrocolpopexie at the Kantonsspital Aarau in a prospective cross-sectional study.

Laparoscopic sacrocolpopexy techniques involving the dissection of the presacral space can compromise fibers of the superior hypogastric plexus. This can contribute to postoperative problems such as incomplete voiding, defecatory dysfunction, pain, and sensory problems. In 2010, the Kantonsspital Aarau has implemented a new nerve-sparing laparoscopic sacrocolpopexy technique. This technique has subjectively reduced the prevalence of stool outlet obstructions but this has not been tested systematically yet. The aim of this study is therefore to compare the patients' subjective conditions between these two surgical techniques using the investigator's standard-of-care German pelvic floor questionnaire.

DETAILED DESCRIPTION:
The (pre-) sacral space is characterized by a complex neuroanatomy and surgical intervention in this part of the body is often associated with the dissection of nerve bundels, a procedure which may finally lead to transient defecatory dysfunction. In a earlier study we could show that ~17.8% of patient with laparoscopic sacrocolpopexie developed postoperative constipation within 3-6 months. In november 2010 the Frauenklinik Aarau introduced a novel, nerve-sparing technique of laparoscopic sacrocolpopexie. In this study we assess the pre-and postoperative differences in defecatory dysfunction between the two procedures trough the analysis of our standard of care pelvic floor questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Women affected by symptomatic vault prolapse, who underwent laparoscopic sacrocolpopexy at the KSA
* informed consent

Exclusion Criteria:

* participation in other studies
* Sacrocolpopexie done by Da Vinci Roboter
* Patients who had a conversion to laparotomy perioperatively
* Patients with a recurrence who had to undergo a second surgery
* Patients who had a relaps operation

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: female patients who underwent laparoscopic sacrocolpopexy at the Kantonsspital Aarau
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
the number of de novo or worsened obstructed defecation | 2003-2017
  comparison of the number of de novo or worsened obstructed defecation of a cohort of patients who underwent nerve-sparing laparaoscopic sacrocolpopexy versus patients who underwent non-nerve-sparing laparaoscopic sacrocolpopexy

CONTACTS AND LOCATIONS:
Overall Officials: Dimitri Sarlos, PD Dr. med., Principal Investigator — Kantonsspital Aarau

REFERENCES:
- [Background] Sarlos D, Brandner S, Kots L, Gygax N, Schaer G. Laparoscopic sacrocolpopexy for uterine and post-hysterectomy prolapse: anatomical results, quality of life and perioperative outcome-a prospective study with 101 cases. Int Urogynecol J Pelvic Floor Dysfunct. 2008 Oct;19(10):1415-22. doi: 10.1007/s00192-008-0657-0. Epub 2008 Jun 7. PMID 18536861
- [Background] Shiozawa T, Huebner M, Hirt B, Wallwiener D, Reisenauer C. Nerve-preserving sacrocolpopexy: anatomical study and surgical approach. Eur J Obstet Gynecol Reprod Biol. 2010 Sep;152(1):103-7. doi: 10.1016/j.ejogrb.2010.05.009. Epub 2010 Jun 9. PMID 20542624
- [Background] Cosma S, Menato G, Ceccaroni M, Marchino GL, Petruzzelli P, Volpi E, Benedetto C. Laparoscopic sacropexy and obstructed defecation syndrome: an anatomoclinical study. Int Urogynecol J. 2013 Oct;24(10):1623-30. doi: 10.1007/s00192-013-2077-z. Epub 2013 Mar 29. PMID 23538995
- [Background] Sarlos D, Kots L, Ryu G, Schaer G. Long-term follow-up of laparoscopic sacrocolpopexy. Int Urogynecol J. 2014 Sep;25(9):1207-12. doi: 10.1007/s00192-014-2369-y. Epub 2014 Apr 4. PMID 24700356